CLINICAL TRIAL: NCT00248404
Title: A Phase I/II Study of NB1011 Administered Intravenously by Continuous Infusion in an Every Second Week Regimen With Open-label Continuation in Cancers That Overexpress the Enzyme Thymidylate Synthase
Brief Title: NB1011 Administered by Continuous Infusion in Cancers That Overexpress Thymidylate Synthase (TS)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kiadis Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR-TSC-001; NCT00255736 (obsolete NCT alias)
Record Dates: First submitted 2005-11-03; First posted 2005-11-04 (Estimated); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Tumors
Keywords: colorectal cancer; ovarian cancer; lung cancer; breast cancer; small bowel cancer; Advanced, recurrent, or metastatic solid tumors of any type; TS overexpression confirmed by fresh biopsy (RTPCR); Suitable for experimental monotherapy
MeSH Terms: conditions — Neoplasms; Colorectal Neoplasms; Ovarian Neoplasms; Lung Neoplasms; Breast Neoplasms; Recurrence | interventions — NB1011

INTERVENTIONS:
Drug: NB1011

SUMMARY:
The purpose of this trial is to assess the tolerability and safety of NB1011 in the treatment of patients with cancers that overexpress TS, such as ovarian, gastrointestinal, colorectal, bladder, breast, and lung cancers.

ELIGIBILITY:
Inclusion Criteria:

* Advanced, recurrent, or metastatic solid tumors
* TS overexpression (> 4 by reverse transcription polymerase chain reaction [RT-PCR]) in archival and fresh samples
* Suitable for experimental monotherapy
* Measurable disease

Exclusion Criteria:

* Tumors that cannot be biopsied or with low level of TS expression
* Requirement for concomitant anticancer therapy
* Treatment with another investigational product within 30 days of study entry
* Pregnant or lactating women
* Active or uncontrolled serious bacterial, viral, fungal, or parasitic infection.
* HIV infection
* Clinically apparent meningeal or central nervous system (CNS) metastases or carcinomatous meningitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Estimated)
Dates: Start 2005-09 (Actual); Primary Completion 2007-12-12 (Actual); Study Completion 2007-12-12 (Actual)

PRIMARY OUTCOMES:
Safety/tolerability of NB1011 infusions
Determination of maximum tolerated dose (MTD)

SECONDARY OUTCOMES:
Pharmacokinetics of NB1011 and its metabolite
Clinical activity as per Response Evaluation Criteria in Solid Tumors (RECIST) criteria
Assessment of TS overexpression

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - University of Minnesota, Minneapolis, Minnesota
- Princess Margaret Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Neuteboom ST, Karjian PL, Boyer CR, Beryt M, Pegram M, Wahl GM, Shepard HM. Inhibition of cell growth by NB1011 requires high thymidylate synthase levels and correlates with p53, p21, bax, and GADD45 induction. Mol Cancer Ther. 2002 Apr;1(6):377-84. PMID 12477050
- [Background] Salonga D, Danenberg KD, Johnson M, Metzger R, Groshen S, Tsao-Wei DD, Lenz HJ, Leichman CG, Leichman L, Diasio RB, Danenberg PV. Colorectal tumors responding to 5-fluorouracil have low gene expression levels of dihydropyrimidine dehydrogenase, thymidylate synthase, and thymidine phosphorylase. Clin Cancer Res. 2000 Apr;6(4):1322-7. PMID 10778957
- [Background] Lenz HJ, Leichman CG, Danenberg KD, Danenberg PV, Groshen S, Cohen H, Laine L, Crookes P, Silberman H, Baranda J, Garcia Y, Li J, Leichman L. Thymidylate synthase mRNA level in adenocarcinoma of the stomach: a predictor for primary tumor response and overall survival. J Clin Oncol. 1996 Jan;14(1):176-82. doi: 10.1200/JCO.1996.14.1.176. PMID 8558194
- [Result] Pegram M, Yeon CH, Ku N, Gottlieb C, Sheppard M, Cossum P, John E, Iqbal S, Garcia A, Lenz HJ. Enzyme Catalyzed Therapeutic Activation of NB1011 Selectively Targets Thymidylate Synthase-overexpressing Tumor Cells: Phase I Results. ASCO Meeting, New Orleans, June 4-8, 2004 (abstract 3144)